CLINICAL TRIAL: NCT04023123
Title: The Clinical Significance of Anterior Corneal Striae in Hypotony
Brief Title: Anterior Corneal Striae in Hypotony
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00102744
Record Dates: First submitted 2019-07-11; First posted 2019-07-17 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2019-06

CONDITIONS: Hypotony Ocular; Cornea Folds and Rupture of Bowman's Membrane Both Eyes; Maculopathy
MeSH Terms: conditions — Ocular Hypotension; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anterior Cornea Striae: Eyes with anterior cornea striae present
  Interventions: Other: Ophthalmic imaging
- Hypotony Maculopathy: Eyes with hypotony maculopathy present
  Interventions: Other: Ophthalmic imaging
- Hypotony only: Eyes with intraocular pressure less than 10 without cornea striae and/or maculopathy
  Interventions: Other: Ophthalmic imaging

INTERVENTIONS:
Other: Ophthalmic imaging — Optical coherence tomography Topography Ocular Response Analyzer Optical Biometry Slit lamp photos

SUMMARY:
The goal of this is to evaluate the biomechanical properties of hypotonous eyes with vertical anterior corneal striae and/or hypotony maculopathy compared to hypotonous eyes without striae.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >= 18 years of age
* History of glaucoma
* History of glaucoma surgery
* Intraocular pressure of equal to or less than 10 mm Hg by goldmann applanation

Exclusion Criteria:

* Coexisting ocular disease that may affect ocular biomechanics, including macular disease, corneal transplant, and uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects >= 18 years of age with a history of glaucoma and glaucoma surgery
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Corneal hysteresis | Baseline
  Difference in postoperative corneal hysteresis (measured in mm Hg) by Ocular Response Analyzer, between study arms
Incidence of anterior corneal striae | Baseline
  Frequency of occurrence among all enrolled hypotonous eyes
Incidence of hypotony maculopathy | Baseline
  Frequency of occurrence among all enrolled hypotonous eyes

SECONDARY OUTCOMES:
Axial length | Baseline
  Difference in postoperative axial length between study arms
Corneal thickness | Baseline
  Difference in postoperative corneal thickness between study arms
Corneal curvature | Baseline
  Difference in postoperative diopters of steepest cornea axis, flattest cornea axis and astigmatism between study arms
Corneal resistance factor | Baseline
  Difference in postoperative corneal resistance factor between study arms

CONTACTS AND LOCATIONS:
Overall Officials: Leon Herndon, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No